CLINICAL TRIAL: NCT01650441
Title: OPEN-LABEL, PROSPECTIVE EXPLORATORY STUDY TO ASSESS THE EFFECTS OF FORMOTEROL AND BECLOMETASONE DIPROPIONATE COMBINATION THERAPY USING A DPI DEVICE ON CENTRAL AND PERIPHERAL AIRWAY DIMENSIONS IN ASTHMATIC PATIENTS.
Brief Title: Study to Assess the Effect of the NEXThaler® Device (DPI - Dry Powder Inhaler) on the Central and Peripheral Airway Dimensions in Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Wilfried De Backer, MD PhD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PML_DOC_1102; 2011-003249-16 (EudraCT Number)
Record Dates: First submitted 2012-06-29; First posted 2012-07-26 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
Keywords: Asthma; NEXThaler®; Formoterol; Beclomethasone Dipropionate; Computational Fluid Dynamics; Functional Imaging; Central and Peripheral Airways; Asthma Control Test (ACT™); Asthma Control Questionnaire (ACQ)
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- beclomethasone dipropionate + formoterol fumarate (Experimental): All patients will be treated with the active product. No placebo arm will be used. The active product is a fixed combination containing extra-fine beclometasone dipropionate and formoterol fumarate in a new dry powder inhaler device, NEXThaler® (Chiesi Farmaceutici, Parma, Italy).
  Interventions: Drug: Beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg; Radiation: CT thorax

INTERVENTIONS:
Drug: Beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg — In this trial, patients will take two inhalations of the beclometasone dipropionate 100 µg and formoterol fumarate 6 µg combination therapy (Foster®) using a Dry Powder Inhaler (NEXThaler®) device in the morning and two inhalations in the evening, for a total of 4 inhalations a day (total daily dose: BDP 400 µg / FF 24 µg).
  Other Names: NEXThaler®
Radiation: CT thorax — CT scan of the thorax will be performed at 2 time points: baseline and after 6 months of treatment.
  The CT scan will be performed with low dose radiation using the multi-slice CT scan. Scanning will be performed at Functional Residual Capacity and Total Lung Capacity (2 times 8 sec). The lung volumes will be controlled using adapted spirometry during the CT procedure. The radiation dose will be reduced by reduction of the tube current and voltage. These settings depend on the patients' weight (1mAs/kg). In addition to this there will be an increase in noise factor to further reduce the radiation dose.

SUMMARY:
The objective of this study is to evaluate the effect of the combination of formoterol and beclometasone dipropionate in a dry powder inhaler (NEXThaler®) on central and peripheral airway dimensions in asthmatic patients. Therefore Computational Fluid Dynamics (CFD) will be used. Further more, the effect of this combination therapy on lung function (spirometry, resistance and diffusion), the Asthma Control Test (ACT™) and the Asthma Control Questionnaire (ACQ) will be assessed and the safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate asthma as defined by the current GINA guidelines. Patients can belong to 2 categories:

   Group 1 (n=15 to 20, at least 4 current smokers): Patients not well controlled (partially controlled or uncontrolled according to the GINA guidelines) when using medium daily dose of ICS or medium dose ICS + long acting inhaled 2-agonists (LABA) (for definition please refer to the addendum in section 15) given for at least 6 weeks as large-particle formulation (non extra-fine).

   Group 2 (n=15 to 20, at least 4 current smokers ): Patients well controlled (according to GINA guidelines) when using medium daily dose of ICS + LABA (for definition please refer to the addendum in section 15) given for at least 6 weeks as large-particle formulation (non extra-fine).
2. Male or female patients aged ≥18 years
3. Patients with a documented diagnosis of asthma according to the GINA guidelines
4. Patients with a co-operative attitude and ability to be trained to correctly use the Foster NEXThaler DPI
5. Written informed consent obtained

Exclusion Criteria:

1. Patients treated with extra-fine ICS either alone or with LABA
2. Pregnant or lactating females or females at risk of pregnancy at screening and not willing to use an appropriate contraception method during the study period
3. Inability to carry out pulmonary function testing
4. History of near fatal asthma
5. Hospitalization due to asthma or symptomatic infection of the airways in the previous 8 weeks
6. Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
7. Cancer
8. Current alcohol or drug abuse
9. Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients
10. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
11. Patients who received any investigational new drug within the last 4 weeks prior to the screening visit
12. Patients treated with any non-permitted concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Computational Fluid Dynamics (CFD) | CFD will be performed based on the images of 2 CT thorax scans in a dose reduction protocol (1 CT Thorax taken at baseline and 1 CT Thorax taken after 6 months of treatment with the NEXThaler® device).
  The parameters that will be obtained with the CFD based imaging and used as primary outcome parameters are:
  * Total airway resistance for the segmented airways iRtot
  * Peripheral airway resistance(from 4th bifurcation on) for the segmented airways iRperph
  * Total airway volume for the segmented airways (iVtot)
  * Peripheral airway volume (from the 4th bifurcation on) for the segmented airways (iVperiph)
  * Relative compliance for each lobe (iClobe-rel)
  * Density of the lung parenchyma given per predefined lung zone (Ldens)

SECONDARY OUTCOMES:
Lung function tests | Lung function tests will be performed at screening (visit 1), after 2 week run-in period both pre and post dose (visit 2), after 3 months treatment (visit 5), after 6 months treatment both pre and post dose (visit 8).
  The parameters that will be obtained with the described lung function tests are:
  * Dynamic lung volumes: FEV1, FVC, PEF, MEF75, MEF50, MEF25
  * Static lung volumes: VC, IVC, FRC, TLC
  * Airway resistances: Raw, SGaw
Asthma Control | Asthma control will be monitored at screening (visit 1), after 2 week run-in period (visit 2), after 3 months treatment (visit 5), after 6 months treatment (visit 8).
  Asthma Control will be monitored during the study using 2 different questionnaires: the Asthma Control Test (ACT™) and the Asthma Control Questionnaire (ACQ, both the 6-items and the 7-items test will be used.)
Safety | The safety of the NEXThaler® device will be monitored for the duration of the study, an expected average of 24 weeks.
  During the study the patient will be told to record each day taken medication and any possible comments on the daily diary cards, starting from visit 1. Further more, the patient will be contacted at least once a month (either by phone or a visit in the hospital.)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD PhD, Principal Investigator — University Hospital of Antwerp
Locations (1):
- University Hospital of Antwerp, Edegem (Antwerp), Antwerp, Belgium